CLINICAL TRIAL: NCT05842486
Title: Hematological Response in Patients With Paroxysmal Nocturnal Hemoglobinuria Treated With Anti-C5 Antibody: an External Control Arm Study for Iptacopan Use in Anti-C5 naïve Patients
Acronym: APPEX
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Leeds Cancer Centre at St. James's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CLNP023N12002R
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Real-world cohort: The real-world cohort consists of patients with diagnosis of paroxysmal nocturnal hemoglobinuria and anemia initiating anti-C5 therapy.
  Interventions: Other: Anti-C5 antibody treatment

INTERVENTIONS:
Other: Anti-C5 antibody treatment — Anti-C5 antibody treatment (i.e., eculizumab and ravulizumab)

SUMMARY:
The aim of this non-interventional secondary use of data study is to evaluate hematological response in patients with paroxysmal nocturnal hemoglobinuria and anemia in the 6-month period after initiation of anti-C5 antibody treatment using real-world data obtained from multiple datasets. The results will be used to contextualize results from the APPOINT-PNH (NCT04820530) trial with iptacopan.

ELIGIBILITY:
Inclusion Criteria:

1. Incident users of anti-C5 antibody treatment (i.e., first use of anti-C5 antibody with no evidence of use prior to that)
2. Confirmed clinical diagnosis of PNH (including PNH clone size >10% in RBC percent/white blood cell (WBC) percent)
3. Adult patients ≥18 years of age
4. Baseline Hb <10 g/dL.

Exclusion Criteria:

Patients who met any of the following criteria were not eligible for inclusion.

1. Bone marrow transplantation within one year prior to initiating anti-C5 treatment
2. Hereditary complement deficiency
3. Reticulocyte count <60x10^9/L.
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The real-world cohort consists of patients with diagnosis of paroxysmal nocturnal hemoglobinuria and anemia initiating anti-C5 therapy. Patient data originate from the Hôpital Saint-Louis, France and St. James's University Hospital, Leeds, United Kingdom.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Increase from baseline in hemoglobin | between Day 100 and Day 200
  Increase from baseline in hemoglobin of ≥ 2 g/dL in the absence of transfusions occurring after Day 14 post index date

SECONDARY OUTCOMES:
Hemoglobin Response | between Day 100 and Day 200
  Achieving hemoglobin of ≥ 12 g/dL in the absence of blood transfusions occurring after Day 14 post index date
Transfusion avoidance | Occurrence between Day 15 and Day 200
  Transfusion avoidance (dichotomous endpoint) defined proportion of subjects without transfusions during the initial 6-month treatment period starting from 2 Weeks after index date (i.e., date of first anti-C5 antibody treatment for PNH).

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holt M, Kelly RJ, Fermont JM, Ansari S, Dahlke M, Brindel I, Maafa L, de Fontbrune FS, de Latour RP. Effectiveness of Iptacopan Versus C5 Inhibitors in Complement Inhibitor-Naive Patients With Paroxysmal Nocturnal Haemoglobinuria. EJHaem. 2025 May 20;6(3):e270055. doi: 10.1002/jha2.70055. eCollection 2025 Jun. PMID 40395624